CLINICAL TRIAL: NCT06209424
Title: Non-Invasive Modified Breath Test to Determine Anabolic Sensitivity Across Physical Activity States in Healthy Young Adults
Brief Title: Modified Breath Test to Determine Anabolic Sensitivity Across Physical Activity States
Acronym: BTLP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Toronto (Other)
Responsible Party: Principal Investigator, Daniel Moore, Principal Investigator, University of Toronto
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 00044918
Record Dates: First submitted 2024-01-05; First posted 2024-01-17 (Actual); Last update posted 2024-01-17 (Actual); Status verified 2024-01

CONDITIONS: Resistance Exercise; Physical Inactivity; Amino Acids; Dietary Protein
Keywords: Sex; Step-Reduction; Habitual Activity; Protein Metabolism; Resistance Exercise; Stable Isotopes; Anabolic Sensitivity
MeSH Terms: conditions — Sedentary Behavior; Coitus | interventions — Resistance Training

STUDY DESIGN:
Intervention Model Description: Randomized Counter-Balanced Crossover Design
  Following familiarization, participants will be split into an in-person phase, consisting of a habitual rest and subsequent whole-body resistance exercise metabolic trials, and an at-home phase, which includes a habitual rest followed by a step-reduction metabolic trial. Participants will be randomized through a counterbalanced approach to either start with the in-person or at-home phases of our study as outlined below. Participants will be grouped by sex to ensure the same number of individuals from both males and females will undergo the in-person or at-home phases first
Masking Description: Participants will be randomized to either begin their participation with the "at-home" or "in-person" phase of the study. There is no need to conceal the randomization as this study is not blinded - this does not affect our outcome as we are looking at physiological changes with feeding.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- In-Person Phase (Active Comparator): Habitual Activity + Resistance Exercise Metabolic Trials
  Interventions: Behavioral: Habitual Activity; Behavioral: Resistance Exercise
- At-Home Phase (Active Comparator): Habitual Activity + Step-Reduction Metabolic Trials
  Interventions: Behavioral: Habitual Activity; Behavioral: Step-Reduction

INTERVENTIONS:
Behavioral: Habitual Activity — Participants will maintain habitual levels of physical activity (inclusive of structured physical activity).
  Other Names: Free-Living Activity
Behavioral: Step-Reduction — Participants will be required to reduce their daily step-counts to <2,000 steps/day. Further, they will be required to refrain from structured physical activity.
  Other Names: Reduced Physical Activity
  Arms: At-Home Phase
Behavioral: Resistance Exercise — Participants will undergo a 50-minute resistance exercise protocol, which includes multiple sets of different exercises using weights. Each set will consist of 10 repetitions at 75% of their 1 repetition maximum (1RM). The exercises include bench press superset with lat pulldowns, overhead press superset with seated cable rows, leg press, and leg extensions with 90s rest in between sets. Before the exercise protocol, there will be a standardized 10-minute warm-up that involves cycling, leg swings, arm circles, bodyweight squats, and bench push-ups
  Other Names: Full-Body Resistance Exercise
  Arms: In-Person Phase

SUMMARY:
Developing tools to detect when our bodies are more resistant towards protein synthesis is valuable for identification of when someone may be at risk of losing body or muscle mass such as with aging or certain diseases. The current study aims to refine our previous breath test method to be more effective at measuring changes in how the body processes protein in different situations, such as resting, reducing physical activity, and doing resistance exercise. We hypothesize that using a lower amount of dietary amino acids in our breath test will be effective at detecting lower amounts of amino acids used after exercise, and a greater amount with step reduction compared to normal activity levels

DETAILED DESCRIPTION:
Maintaining high-quality and abundant lean body mass (LBM) is crucial for growth, health, and performance across all ages, sexes, and activity levels. Body protein, including skeletal muscle, undergoes constant turnover, breaking down old and damaged proteins and using dietary amino acids (AA) to synthesize new proteins, especially after resistance exercise. Unused AA are oxidized for energy and excreted as carbon dioxide (CO2). Studying the proportion of AA used for protein synthesis versus energy production provides insights into acute growth of LBM after a meal in different physiological states (e.g., at rest or exercise). Stable isotope tracers, commonly administered intravenously, are used in protein metabolism research to examine the effects of nutrition and exercise on protein turnover. However, this method may not be feasible for vulnerable populations.

While exercise has been shown to enhance anabolic sensitivity (i.e., greater utilization of dietary AA for protein synthesis), step-reduction leads to fed-state anabolic resistance (I.e., reduced utilization of dietary AA for protein synthesis). Indeed, reduced habitual activity, whether mild or severe, leads to fed-state anabolic resistance, reducing the muscle protein synthesis (MPS) response to amino acids. For instance, one week of reduced daily steps (~1,192 steps/day) decreased MPS rates by approximately 27% in young males who habitually reach ~10,000 steps/day, i.e., a ~75% reduction from habitual.

Therefore, developing metabolic tools to detect anabolic resistance before muscle mass loss occurs would be valuable for both treatment and prevention of age-related muscle loss. Recently, our laboratory demonstrated the effectiveness of a non-invasive stable isotope "breath test" to detect increased anabolic sensitivity in males after resistance exercise. This study, in addition to ongoing metabolic trials in our lab, utilized a protein dose of 0.25g/kg which has been shown to maximize the rate of myofibrillar protein synthesis and to support whole-body protein synthesis. However, this dose may not adequately distinguish between more subtle changes in anabolic sensitivity. Further, a lower protein dose may reduce the duration for which breath samples would need to be collected, which would minimize participant burden and time commitment going forward.

Therefore, the present project will use previously established 'breath test' methodology but with a lower protein dose to assess the following objectives:

1. To investigate whether the 'optimized' non-invasive breath test can detect changes in anabolic sensitivity (i.e., leucine oxidation) across varying physiological states (I.e., rest, step-reduction, whole-body resistance exercise) after feeding, in young healthy adults.
2. To assess the reproducibility, and day-to-day variability of our breath test during habitual activity in both an at-home and a controlled laboratory setting

ELIGIBILITY:
Inclusion Criteria:

* Healthy young (age: 18-35 years)
* BMI between normal to overweight (18.5-29.9 kg/m2)
* if oral contraceptive (OC) user, must be on monophasic OCs for at least 3 months prior to study
* if non-OC user, then must have regular menstrual cycles (length: 25-35 days) for at least 3 months prior to study and at least 6 months off of OCs

Exclusion Criteria:

* Chronic disease diagnosis (cardiovascular, thyroid, diabetes)
* Current or recent remission of cancer
* Regular use of NSAID (except low-dose aspirin), anticoagulants
* Use of prescription drugs that would impact muscle protein synthesis (e.g., Statins, Lithium, ADHD medication, etc..)
* Insertion of intrauterine device (IUD) - exception: copper
* Smoking
* Use of illicit drugs (growth hormones, testosterone)

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Estimated)
Dates: Start 2024-01-15 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
Exogenous Leucine Oxidation (umol/kg) | 5 hours
  Exogenous Leucine Oxidation determined from breath 13CCO2 enrichment. Breath samples will be collected every 20-30min after test drink ingestion to determine breath 13CO2 enrichment. Total leucine oxidation will be determined from the area under the 13CO2 enrichment by time curve.
Net Leucine Retention (umol/kg) | 5 hours
  Whole-Body Net Leucine Retention determined from the difference between exogenous leucine oxidation and leucine ingestion the 6 hour measurement period.

OTHER OUTCOMES:
Feeling and Felt Arousal (Likert Scale) | 6 days (during at-home phase)
  Feeling and felt arousal will be assessed 3-times a day in conjunction with mealtimes (i.e., breakfast, lunch, dinner) to understand whether acute periods of inactivity are sufficient to induce changes in activation and arousal states in otherwise healthy active individuals

CONTACTS AND LOCATIONS:
Overall Officials: Ines Kortebi, MSc, Study Director — University of Toronto; Hugo JW Fung, PhD (c), Study Chair — University of Toronto; Daniel R Moore, PhD, Principal Investigator — University of Toronto
Locations (1):
- Goldring Centre for High Performance Sport at the University of Toronto, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No